CLINICAL TRIAL: NCT04591041
Title: HoloSIM: The Way Forward in Complex Crisis Training
Brief Title: HoloSIM: Mixed Reality Medical Student Training in Complex Crisis Scenarios
Acronym: HoloSIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Julian Wiegelmann, Anesthesiologist, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUN-2124
Record Dates: First submitted 2020-09-02; First posted 2020-10-19 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Simulation of Physical Illness; Educational Problems
Keywords: Mixed Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training by Mixed Reality Simulation (Experimental)
  Interventions: Device: HoloSIM Software via Hololens 2
- Training by Mannequin Based Simulation (Active Comparator)
  Interventions: Other: Training by Mannequin Based Simulation

INTERVENTIONS:
Device: HoloSIM Software via Hololens 2 — Medical students will train via a mixed reality simulated crisis scenario using the HoloSIM software on the Microsoft Hololens 2
  Arms: Training by Mixed Reality Simulation
Other: Training by Mannequin Based Simulation — Medical students will train a via traditional mannequin based medical crisis scenario
  Arms: Training by Mannequin Based Simulation

SUMMARY:
In this study, Investigators will test a mixed reality software platform to improve and help for teaching and assessment of anesthesia crisis management among medical students.

ELIGIBILITY:
Inclusion Criteria:

* University of Toronto Medical student volunteers

Exclusion Criteria:

* Unwilling to enter the study
* Deficit of vision or hearing incompatible with Microsoft Hololens 2 use

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Anaphylaxis Checklist of Core Decision Making Steps | one week post exposure
  Expert consensus based checklists of critical scenario actions on a mannequin based crisis scenario. Student scenario performance graded from 0 to 45, with higher scores representing a better performance.

SECONDARY OUTCOMES:
Usability Score | Immediately after exposure
  Likert scale (5 point) based assessment of software usability. Higher scores on a scale of 1 to 5 represent a better software system usability.
Learning Satisfaction Score | Immediately after exposure
  Likert scale (5 point) based assessment of learning satisfaction. Higher scores on a scale of 1 to 5 represent a greater degree of learning satisfaction.
Time required to complete critical crisis related tasks | one week post exposure
  Measured time until critical scenario management events occur

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No